CLINICAL TRIAL: NCT00209287
Title: Study of Histological Modifications, of Pro-apoptotic Effects and of Modifications in Apoptosis Regulators Observed After Stopping 5-ASA Treatment in Patients With Inactive Ulcerative Colitis (Clinical and Endoscopic Remission) Taking 5-ASA
Brief Title: Study of Effects and of Modifications in Apoptosis Regulators Observed After Stopping 5-ASA Treatment in Patients With Inactive Ulcerative Colitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment problematic
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Mesalazine 2004-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis for Maintenance of Remission
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Observe patients with inactive ulcerative colitis — Observe patients with inactive ulcerative colitis

SUMMARY:
Male or female, 18 years of age or older. Ulcerative Colitis described according usual criteria, diagnosed for at least 1 year. Oral maintenance treatment with 5-aminosalicylic acid (5-ASA) only for at least 3 months with a dosage of 2 to 3 g/day. Clinical remission for at least 3 months (Mayo Clinic score) and endoscopic remission (endoscopic score of Mayo Clinic) at the inclusion. Signed informed consent form.

DETAILED DESCRIPTION:
Inclusion Criteria:

* Male or female, 18 years of age or older.
* Ulcerative colitis described according to usual criteria, diagnosed for at least 1 year.
* Oral maintenance treatment with 5-aminosalicylic acid (5-ASA) only for at least 3 months with a dosage of 2 to 3 g/day.
* Clinical remission for at least 3 months (Mayo Clinic score) and endoscopic remission (endoscopic score of Mayo Clinic) at inclusion.
* Signed informed consent form.

Exclusion Criteria:

* Patients allergic to aspirin or salicylates derivatives
* Patients taking the following treatments during the study will be excluded: corticosteroids (oral or rectal route), use of NSAID or Aspirin, any form of sulfasalazine, mesalazine or 4-ASA.
* Patients with known significant hepatic or known function abnormalities and/or creatine clearance ≤ 80 ml/min.
* Patients with history or physical examination findings indicative of active alcohol or drug abuse.
* Women who are pregnant or nursing.
* Patients with a history of disease, including mental/emotional disorder that would interfere with their participation in the study.
* Patients who participated in another clinical study in the last 3 months.
* Patients who are unable to comply with the requirements of the protocol
* Female of childbearing potential without efficacious contraception.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older.
* Ulcerative colitis described according to usual criteria, diagnosed for at least 1 year.
* Oral maintenance treatment with 5-ASA only for at least 3 months with a dosage of 2 to 3 g/day.
* Clinical remission for at least 3 months (Mayo Clinic score) and endoscopic remission (endoscopic score of Mayo Clinic) at inclusion.
* Signed informed consent form.

Exclusion Criteria:

* Patients allergic to aspirin or salicylates derivatives
* Patients taking the following treatments during the study will be excluded: corticosteroids (oral or rectal route), use of NSAID or Aspirin, any form of sulfasalazine, mesalazine or 4-ASA.
* Patients with known significant hepatic or known function abnormalities and/or creatine clearance ≤ 80 ml/min.
* Patients with history or physical examination findings indicative of active alcohol or drug abuse.
* Women who are pregnant or nursing.
* Patients with a history of disease, including mental/emotional disorder that would interfere with their participation in the study.
* Patients who participated in another clinical study in the last 3 months.
* Patients who are unable to comply with the requirements of the protocol
* Female of childbearing potential without efficacious contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-06; Primary Completion 2006-12 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change between rectal biopsies performed at D1 and D28 of proliferative index | Its aim was to study histological modifications after Pentasa was stopped in non-active ulcerative colitis.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Hôpital Saint Antoine, Service d'hépato-Gastroentérologie, Paris, France